CLINICAL TRIAL: NCT04549610
Title: The Effect of β-hydroxy-β-methylbutyrate Supplementation on Muscle Damage Induced by Resistance Exercise
Brief Title: HMB and Exercise-induced Muscle Damage
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Collaborators: Escola de Educação Física e Esporte da Universidade de São Paulo (Brazil) - Parallel sponsor of the research (Unknown); National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Krzysztof Durkalec-Michalski, Prof Dr hab., PhD, Poznan University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ULS2020.001
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Supplementation; Sport; Sports Nutrition; Muscle Damage; Recovery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMB supplementation (Experimental): The experimental procedure for each participant in this group includes a one week HMB supplementation.
  HMB will be administered in the form of blinded capsules containing 0.5 g HMB per capsule. The capsules will be ingested with at least 250 mL of water. Each athlete will ingest 8 capsules (4 x 2 capsules) of HMB in a split dose per day. On training days the supplements will be taken in the morning (2 capsules), 1.5 hours before training session (2 capsules), immediately after training (2 capsules) and before sleep (2 capsules). On rest days the supplements will be taken in the morning (2 capsules), around midday (2 capsules), in the afternoon (2 capsules) and before bedtime (2 capsules) at possibly similar (approx. 4 hours) intervals during the day.
  Interventions: Dietary Supplement: HMB supplementation
- Placebo treatment (Placebo Comparator): The experimental procedure for each participant in this group includes a one-week placebo (PLA) administration. PLA (corn starch) will be placed in the blinded capsules form. PLA will be ingested with at least 250 mL of water. Each participant in this group will ingest 8 placebo capsules a day. On training days the PLA capsules will be taken in the morning (2 capsules), 1.5 hours before training session (2 capsules), immediately after training (2 capsules) and before sleep (2 capsules). On rest days the supplements will be taken in the morning (2 capsules), around midday (2 capsules), in the afternoon (2 capsules) and before bedtime (2 capsules) at possibly similar (approx. 4 hours) intervals.
  Interventions: Dietary Supplement: Placebo treatment

INTERVENTIONS:
Dietary Supplement: HMB supplementation — Group taking oral HMB supplementation in a blinded capsule form.
  Arms: HMB supplementation
Dietary Supplement: Placebo treatment — Group taking oral supplementation with placebo (corn starch) in a blinded capsule form.
  Arms: Placebo treatment

SUMMARY:
The study aims at assessing the influence of β-hydroxy-β-methylbutyrate (HMB) supplementation (4.0 g/day) supplemented for 7 days in a group of speed-strength trained individuals on lower-body strength performance, selected muscle histological, molecular and blood markers of muscle recovery in response to resistance exercise-induced muscle damage.

DETAILED DESCRIPTION:
The main aim of the project is to assess the effects of seven days of HMB (4.0 g/day) or Placebo (PLA) supplementation on lower body strength performance, and functional, histological, clinical and molecular markers of muscle recovery after an acute resistance exercise session.

The study is a double-blind, randomized, placebo-controlled, parallel trial. 30 male participants will be divided randomly into two parallel groups: One group receiving 4.0 g/day HMB and the second group receiving PLA. Supplementation period (HMB or PLA) will be seven days (five days before and two days after muscle damage induced by an acute resistance training session). Food intake during the intervention will be assessed with the use of a food diary.

Before the start of the experimental protocol, the participants will be familiarized with all tests and procedures.

During the first visit, participants will be assessed for their anthropometric characteristics, and baseline blood samples will be collected for the analysis of the activity of muscle damage markers [creatine kinase (CK) and lactate dehydrogenase (LDH)]. We will then carry out the evaluation of the maximal voluntary isometric contraction (MVIC; performed in a Biodex isokinetic dynamometer), lower body maximum dynamic strength (1RM) for squat, leg press, and leg extension exercises. The participants will then return to the laboratory to repeat the same tests and confirm the obtained results (MVIC and 1RM tests).

On the third day, participants will take part in a resistance training session (RE3sets) to evaluate strength performance. We will monitor the maximum number of repetitions possible in three sets of three exercises (squats, the leg press, and leg extension), until the concentric failure, with a rest interval of two minutes per set. The workload will correspond to 80% of the individual's 1RM).

Participants will then spend five to seven days without any leg strength/power training, in order to facilitate effective recovery prior to the next main resistance exercises training (RE5sets), which will be designed to induce muscle damage. Furthermore, HMB or PLA supplementation will commence five days before RE5sets, and continue for 48 hours after RE5sets.

Before the RE5sets, a muscle biopsy will be done in the vastus lateralis for morphological analysis of the sarcomere integrity (histological analysis) and molecular testing (e.g. selected protein kinase activity (e.g. AKTser473, mTORSer2448, p70S7K1Thr389, 4E-BP1Ser65/Thr70, 4EBP1Thr37/46); muscle cholesterol, and mevalonate content). Blood samples will also be collected. After the biopsy, participants will carry out exercises similar to those performed in the preliminary studies, but will do 5 sets per exercise until concentric failure with a 2-min resting interval between sets and load corresponding to 80% of the participant's 1RM.

24 hours after the end of RE5sets, blood samples will be taken and the evaluation of the MVIC will be performed. 24 hours later (48 hours after the RE5sets), a muscle biopsy (for histological and molecular testing) will be conducted, and blood samples will be collected. Furthermore, the MVIC and RE3sets will also be measured.

Collected data will be compared between groups and times using mixed models (proc mixed, SAS v.9.3) followed by multiple comparisons of a hypothesis-driven single degree of freedom contrast analysis. The sample size was estimated at 24 in total, assuming an intra- and inter-subject interaction model, alpha level of 5%, power (1-β) of 0.8 and effect size 0.3 (small) (G*Power v.3.9.1.2). We will recruit a slightly larger number of participants (n = 30) to allow for the likely dropouts that will occur throughout the study. The level of significance adopted will be p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent from all participants before the study
* a current medical clearance to practice sports,
* training experience: at least 1 year strength training programs that include lower limbs,
* minimum of 3 workout sessions (strength/resistance training) a week,
* protein intake in customary diet and during the study protocol > 1.6g / kg of body mass per day,
* individual maximum strength greater than 2.5 times the body weight for the 1RM test in the leg-press.

Exclusion Criteria:

* current injury,
* any health-related contraindication,
* declared general feeling of being unwell,
* unwilling to follow the study protocol,
* serious disease or metabolic problems,
* intake of creatine, caffeine or beta-alanine, or other ergogenic supplements 3 months before the beginning of the study,
* history of anabolic androgenic steroids or drugs use that may interfere with muscle mass control (eg, corticosteroids), or affect physical performance,
* smoking and tobacco use,
* presence of infectious disease in the previous 4 weeks of the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the maximum voluntary isometric contraction (MVIC) after supplementation and exercises-induced muscle damage | Baseline, 24 hours and 48 hours after the end of exercises-induced muscle damage
  Maximum voluntary isometric contraction (MVIC) torque (Nm)

SECONDARY OUTCOMES:
Change in the histological sarcomere integrity (after biopsy of the vastus lateralis muscle samples) after supplementation and exercises-induced muscle damage | Baseline, 24 hours and 48 hours after the end of exercises-induced muscle damage
  The disruption of the Z-line areas and the total visible fiber area in muscle fibers (%)
Change in the molecular potential (after biopsy of the vastus lateralis muscle samples) after supplementation and exercises-induced muscle damage | Baseline, 24 hours and 48 hours after the end of exercises-induced muscle damage
  AKTser473, mTORSer2448, p70S7K1Thr389, 4E-BP1Ser65/Thr70, and 4EBP1Thr37/46 kinase activity (optical density)
Change in the muscle cholesterol and mevalonate content (in the vastus lateralis muscle samples) after supplementation and exercises-induced muscle damage | Baseline, 24 hours and 48 hours after the end of exercises-induced muscle damage
  Muscle cholesterol and mevalonate content (units)
Changes in creatine kinase (CK) and lactate dehydrogenase (LDH) activity (IU) in blood after supplementation and exercises-induced muscle damage | Baseline, 24 hours and 48 hours after the end of exercises-induced muscle damage
  CK and LDH activity (IU)
Change in the strength performance results (at 80% of the individual's 1RM) in three resistance exercises (squats, the leg press, and leg extension) before and after supplementation and exercises-induced muscle damage | Baseline and 48 hours after the end of exercises-induced muscle damage
  Number of repetitions in each sets of squats, the leg press, and leg extension (reps)

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme G Artioli, Prof., PhD, Study Chair — Applied Physiology & Nutrition Research Group, University of Sao Paulo. Sao Paulo, SP. Brazil.; Krzysztof Durkalec-Michalski, Dr hab., PhD, Principal Investigator — Department of Sports Dietetics, Poznan University of Physical Education, Poznań, Poland
Locations (1):
- Escola de Educação Física e Esporte da USP / School of Physical Education and Sport - USP., São Paulo, São Paulo - SP, Brazil

IPD SHARING:
Plan to Share IPD: Undecided